CLINICAL TRIAL: NCT05746715
Title: A Natural History Study of Preclinical Genetic Creutzfeldt-Jakob Disease (CJD)
Acronym: NHS_CJD
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Eli Sprecher, MD, Head of R&D, Tel-Aviv Sourasky Medical Center
Other Study IDs: 0215-18
Record Dates: First submitted 2023-02-15; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Creutzfeldt-Jakob Disease (CJD)
Keywords: Creutzfeldt-Jakob Disease; Prion disease; E200K mutation
MeSH Terms: conditions — Creutzfeldt-Jakob Syndrome; Prion Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples and cerebral spinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- genetic Creutzfeldt-Jakob Disease (CJD) patients: A group of patients diagnosed with CJD, who are carriers of E200K mutation in the PRNP gene (gCJD)
- Healthy first degree relatives: A group of first-degree healthy relatives (HR) (both carriers and non-carriers of the E200K mutation in the PRNP gene) of patients diagnosed with gCJD.

SUMMARY:
Creutzfeldt-Jakob Disease (CJD) is the most common prion disease in humans causing a rapidly progressive neurological decline and dementia and is invariably fatal. The familial forms (genetic CJD, gCJD) are caused by mutations in the PRNP gene encoding for the prion protein (PrP). In Israel, there is a large cluster of gCJD cases, carriers of an E200K mutation in the PRNP gene, and therefore the largest population of at-risk individuals in the world. The mutation is not necessarily sufficient for the formation and accumulation of the pathological prion protein (PrPsc), suggesting that other, genetic and non-genetic factors affect the age at symptoms onset. Here we present the protocol of a cross-sectional and longitudinal natural history study of gCJD patients and first-degree relatives of gCJD patients, aiming to identify biological markers of preclinical CJD and risk factors for phenoconversion.

The study includes two groups: Patients diagnosed with gCJD, and first-degree healthy relatives (both carriers and non-carriers of the E200K mutation in the PRNP gene) of patients diagnosed with gCJD. At baseline, and at the end of every year (for 4 years), healthy participants are invited for an "in-depth" visit, which includes a clinical evaluation, blood and urine collection, gait assessment, brain MRI, lumbar puncture, and Polysomnography sleep lab (PSG). At 6 months from baseline, and then halfway through each year, participants are invited for a "brief" visit, which includes a clinical evaluation, short cognitive assessment, and blood and urine collection. gCJD patients will be invited for one "in-depth" visit, similar to the baseline visit of healthy relatives.

ELIGIBILITY:
Inclusion Criteria:

* First--degree relative of an E200K gCJD patient.
* Age 50 years or older at baseline.
* Willingness to undergo genetic testing.
* Ability to provide written informed consent under GCP, ICH, and local regulations.
* Willingness and ability to comply with scheduled visits, required study procedures, and laboratory tests.

Exclusion Criteria:

* a clinical diagnosis of CJD

  * Any other medical or psychiatric condition or laboratory abnormality, which in the opinion of the investigator might preclude participation.
  * Previously obtained MRI scan with evidence of clinically significant neurological disorder other than CJD.
  * Current anticoagulant treatment (e.g Non-vitamin K Antagonist Oral Anticoagulants (NOACs), Warfarin, Low Molecular weight Heparin) that might preclude safe completion of LP.
  * Conditions that preclude the safe performance of LP, such as severe lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
  * Conditions that preclude the safe performance of MRI scannings such as subjects who have a pacemaker, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin, or body, or any other known contra-indication for MRI.
  * Active malignant disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of patients diagnosed with CJD, who are carriers of E200K mutation in the PRNP gene (gCJD), and a group of first-degree healthy relatives (HR) (both carriers and non-carriers of the E200K mutation in the PRNP gene) of patients diagnosed with gCJD.
Sampling Method: Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Existence of pathological Prion Protein (PrP) in CSF of mutation carriers | 8 years
  CSF fluid obtained through yearly lumbar puncture of healthy relatives will be explored for the existence of PrP using RTQuic

SECONDARY OUTCOMES:
Changes in Diffusion Tensor Imaging collected using yearly MRI scans in healthy relatives | 8 years
  Analysis of Diffusion Tensor Imaging (DTI) is expected to reveal lower diffusivity and higher fraction anisotropy in prodromal gCJD

CONTACTS AND LOCATIONS:
Overall Officials: Noa Bregman, MD, Principal Investigator — Tel Aviv Medical Center
Locations (1):
- Cognitive Neurology Unit, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omer N, Droby A, Silbak R, Trablus N, Bar David A, Shiner T, Alcalay Y, Alcalay R, Nathan T, Thaler A, Mirelman A, Gana Weisz M, Goldstein O, Glinka T, Orr-Urtreger A, Giladi N, Bregman N. White matter abnormalities in healthy E200K carriers may serve as an early biomarker for genetic Creutzfeldt-Jakob disease (gCJD). J Neurol Neurosurg Psychiatry. 2025 Mar 13;96(3):226-230. doi: 10.1136/jnnp-2024-333751. PMID 39084863
- [Derived] Bregman N, Shiner T, Kave G, Alcalay R, Gana-Weisz M, Goldstein O, Glinka T, Aizenstein O, Bashat DB, Alcalay Y, Mirelman A, Thaler A, Giladi N, Omer N. The natural history study of preclinical genetic Creutzfeldt-Jakob Disease (CJD): a prospective longitudinal study protocol. BMC Neurol. 2023 Apr 14;23(1):151. doi: 10.1186/s12883-023-03193-8. PMID 37069531